CLINICAL TRIAL: NCT01982019
Title: Determination of Serum Levels of the Orexigenic Neuropeptide 26RFa in Obese Female Patients With or Without Diabetes. Influence of Bariatric Surgery
Brief Title: Influence of Bariatric Surgery on Serum Levels of 26RFa
Acronym: RFa-Ba-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/129/HP
Record Dates: First submitted 2013-10-16; First posted 2013-11-13 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Diabetes; Obesity
Keywords: 26RFa; sleeve gastrectomy; diabetes; obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Obese patients with type 2 diabetes (Other): Meal test taking and hormones measure including 26RFa
  Interventions: Behavioral: Meal test taking and hormones measure including 26RFa
- Obese patients witout diabetes (Other): Meal test taking and hormones measure including 26RFa
  Interventions: Behavioral: Meal test taking and hormones measure including 26RFa
- healthy volonteers (Other): Meal test taking and hormones measure including 26RFa
  Interventions: Behavioral: Meal test taking and hormones measure including 26RFa

INTERVENTIONS:
Behavioral: Meal test taking and hormones measure including 26RFa — Meal test taking and blood sampling for the measure of 26RFa and classical hormones implicated in glucose control and obesity

SUMMARY:
The 26RFa was recently discovered in the hypothalamus. In rodents it seems to be related to glucose metabolism and obesity. However, no data exists in obese patients or in patients with diabetes. Thus, the investigators planned to dose 26RFa level in obese patients before and after a sleeve gastrectomy in order to study the effect of a weight loss on its levels. The investigators will also dose 26RFa concentrations in obese patients with type 2 diabetes and in healthy volunteers with normal weight. Comparison of these different groups will permit us to better understand the 26RFa involvement in glucose concentration regulation and in obesity.

DETAILED DESCRIPTION:
The 26RFa is an orexigenic neuropeptide of the Rfamides family, localized in two hypothalamic nuclei. Its increase induced obesity and it is elevated in obese rodents. In addition, in human, it is elevated in anorexic patients. However, no data exists in obese patients or in patients with diabetes. Thus, the investigators planned to measure 26RFa level in obese patients before and after a sleeve gastrectomy in order to study the effect of a weight loss on its levels. The investigators will also dose 26RFa concentrations in obese patients with type 2 diabetes and in healthy volunteers with normal weight. Comparison of these different groups will permit us to better understand the 26RFa involvement in glucose concentration regulation and in obesity.

The investigators will also measure other hormones known to have a major role in glucose metabolism and obesity (ie. insulin, adiponectin).

A meal test will be given to the volunteers in order to study the kinetics' of these molecules during and after food intake.

ELIGIBILITY:
1. Patients :

   1. Inclusion Criteria:

      * Obese patients (with or without type 2 diabetes) with a planned sleeve gastrectomy
   2. Exclusion Criteria:

      * HbA1c >11 %.
2. Healthy volunteers :

   1. Inclusion Criteria:

      * 20 ≤ BMI ≤ 25 kg/m²,
      * with no treatment that may influence the glycemic control,
      * normal electrocardiogram,
      * no disturbance of the following blood tests: CBC, serum electrolytes, glucose,
      * negative serology of HIV, hepatitis B and C,
      * does not participate at another clinical trial in the last 3 months
   2. Exclusion Criteria:

      * severe medical or surgical history, particularly endocrine or cardiac,
      * oedema syndrome,
      * hypertension.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Serum 26RFa levels | About 1 month before a sleeve gastrectomy
  Serum 26RFa levels will be measured in fasting conditions before a sleeve gastrectomy in obese patients with or without diabetes.

SECONDARY OUTCOMES:
Kinetics of 26RFa levels during a test meal | Before (about 1 month) and after a sleeve gastrectomy (D30 and D180), during a test meal (T0, T30, T60, T90, T120, T150 and T180 )
  levels of 26RFa levels will be measured during a meal test before and after a sleeve gastrectomy in obese patients with or without diabetes, and once a time in healthy volunteers.
kinetics of classical hormones implicated in glucose control and obesity | Before (about 1 month) and after a sleeve gastrectomy (D30 and D180), during a test meal (T0, T30, T60, T90, T120, T150 and T180 )
  levels of classical hormones implicated in glucose control and obesity will be measured during a meal test before and after a sleeve gastrectomy in obese patients with or without diabetes, and once a time in healthy volunteers.
Levels of 26RFa and classical hormones implicated in glucose control and obesity just after a sleeve gastrectomy | at D3 after a sleeve gastrectomy
  Levels of 26RFa and classical hormones implicated in glucose control and obesity just after a sleeve gastrectomy (D3) in obese patients with or without diabetes.
score of satiety | Before (about 1 month) and after a sleeve gastrectomy (D3, D30 and D180)
  Score satiety will be calculated using a questionary before and after a sleeve gastrectomy : once a time at D3, and at T0, T90 and T180 during a meal test at D30 and D180, in obese patients with or without diabetes. It will be also calculated in healthy volunteers at T0, T90 and T180 during a test meal.

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan Prevost, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- University Hospital Rouen, Rouen, Haute Normandie, France

REFERENCES:
- [Derived] Khiar H, Leveque E, Lopez AG, Moreau-Grange L, Richard L, Brunel V, Perdrix A, Takhlidjt S, Devere M, Tavolacci MP, Houivet E, Huet E, Degrimaudet B, Travers C, Leprince J, Picot M, Chartrel N, Prevost G. Serum levels of the incretin-like peptide 26RFa are diminished in women living with obesity and diabetes and restored after sleeve gastrectomy: Results from the prospective pilot RFa-Ba-S study. Diabetes Obes Metab. 2024 Dec;26(12):5556-5568. doi: 10.1111/dom.15871. Epub 2024 Sep 30. PMID 39350486